CLINICAL TRIAL: NCT03068091
Title: Assessment of Lung Movement With CT in Healthy Subjects and Patients With ILD
Brief Title: Assessment of Lung Movement With Computed Tomography (CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Principal Investigator, Talissa Altes, MD, Professor and Chair of the Department of Radiology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2006114
Record Dates: First submitted 2017-02-25; First posted 2017-03-01 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Intervention Model Description: All participants will undergo CT and pulmonary function testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pulmonary Assessment (Other): All participants will undergo a Chest CT scan and pulmonary function testing
  Interventions: Device: Chest CT; Diagnostic Test: Pulmonary Function Testing

INTERVENTIONS:
Device: Chest CT — Inspiration and expiration chest CT
Diagnostic Test: Pulmonary Function Testing — Measure lung function

SUMMARY:
The purpose of this study is to determine whether patient with ILD have altered lung compliance on chest CT before they have macroscopic structural changes on CT.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a group of lung disorders in which the lung tissues become inflamed and then damaged. Idiopathic Pulmonary Fibrosis (IPF) is one of the subtypes of ILD which has characteristic histological and CT features. It is well known that microscopic fibrosis occurs in the lungs of IPF patients well before the structural changes of fibrosis become apparent on CT. By combining sophisticated image analysis with CT scans obtained at full inspiration and full expiration, it may be possible to detect earlier changes of IPF than currently possible by looking at macro structural features alone. With the recent development of new therapeutics for IPF, early detection of the disease and improved monitoring of treatment efficacy will become important. Using CT to assess regional lung compliance has the potential to become an easily translated clinical tool.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ILD: Subjects must have a physician diagnosis of ILD and be in stable pulmonary condition at the time of the CT
* Healthy subjects: Subjects must have no history of pulmonary disease and smoked less than 100 cigarettes in their lifetime

Exclusion Criteria:

* Subjects less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talissa Altes, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the sponsor

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulmonary Assessment
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pulmonary Assessment
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Lung Motion as Assessed by CT
Description: A computer algorithm will compare the inspiration and expiration CT scans to determine regional lung motion.
Time Frame: Study visit 1 of a single visit study
Population: A total of 9 IPF subjects and 13 control subject had CT scans that could be analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Pulmonary Assessment: All participants underwent a Chest CT scan and pulmonary function testing
  Chest CT: Inspiration and expiration chest CT
  Pulmonary Function Testing: Measure lung function
Arm/Group | Pulmonary Assessment
Number analyzed (Participants) | 22
Liters
  Lung Volume Inspiration, IPF: number analyzed (Participants) | 9
  Lung Volume Inspiration, IPF | 4.07 (0.98)
  Lung Volume Inspiration, Control: number analyzed (Participants) | 13
  Lung Volume Inspiration, Control | 5.56 (0.9)
  Lung Volume Expiration, IPF: number analyzed (Participants) | 9
  Lung Volume Expiration, IPF | 1.82 (0.30)
  Lung Volume Expiration, Control: number analyzed (Participants) | 13
  Lung Volume Expiration, Control | 2.46 (0.56)

2. Secondary Outcome: Lung Motion: Lobar Strain Which is a Ratio
Description: Lobar strain (S): the volumetric strain of each lobe i [i = Right Upper (RU), Right Lower (RL), Left Lower (LL), and Left Upper (LU)] as the difference in lobe volume between the expanded and contracted states, normalized by the lobe volume in the expanded state
Time Frame: Study visit 1 of a single visit study
Population: 9 idiopathic pulmonary fibrosis (IPF) and 13 control subjects (N=22) had CT's that were able to be analyzed for lobar strain (lung motion).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Pulmonary Assessment
Number analyzed (Participants) | 22
Ratio
  IPF: number analyzed (Participants) | 9
  IPF | 0.37 (0.15)
  Control: number analyzed (Participants) | 13
  Control | 0.39 (0.30)

ADVERSE EVENTS:
Time Frame: This study had a single study visit. Adverse event data was collected at that visit. No follow-up of subjects was performed.
Arm/Group | Pulmonary Assessment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT03068091/Prot_SAP_000.pdf